CLINICAL TRIAL: NCT01891474
Title: An Open, Parallel-group, Randomized, Interventional Study to Compare the Efficacy and Safety of Voice Inception Technique Based U-healthcare Service in Patients With Type 2 Diabetes Mellitus
Brief Title: Efficacy and Safety of Voice Inception Technique Based U-healthcare Service in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Soo Lim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SNUBH_Uhealth2
Record Dates: First submitted 2013-06-28; First posted 2013-07-03 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- U-health care (Experimental): voice inception technique based U-healthcare service
  Interventions: Device: U-health care
- control (No Intervention): conventional treatment

INTERVENTIONS:
Device: U-health care — voice inception technique based U-healthcare service
  Other Names: U-health care group
  Arms: U-health care

SUMMARY:
Ubiquitous healthcare service for elderly patients with type 2 diabetes have been developed and improved glycemic control. However, previous U-healthcare service had some limitations, which needs specific devices to check blood glucose and send it to central system. Voice inception technique based U-healthcare service is expected to improve glycemic control without specific devices.

To evaluate the clinical efficacy of this system, researchers plan to compare the improvement of glycemic control, self-management, and quality of life between U-health care group (intervention) and conventional treatment group (control).

DETAILED DESCRIPTION:
Ubiquitous healthcare for chronic disease such as diabetes is intensively developing field. Nowadays, various methods are tried to find the most effective and easiest way for supplying U-health care.

Here, researchers are going to investigate the efficacy and safety of voice inception technique based U-healthcare service.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* age: 60 ~ 85 yrs
* HbA1c: 7.0%-11.0%
* Basal insulin or premixed insulin user

Exclusion Criteria:

* Type 1 diabetes
* short acting insulin or insulin pump user
* systemic corticosteroid administered within previous 6 months
* history of myocardial ischemia
* Heart failure, New York Heart Association (NYHA) Class II-IV
* Thyroid disease with abnormal thyroid function test
* Anti-obesity drugs or slimming products within previous 3 months
* severe liver or kidney disease

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-08; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Changes of HbA1c | 24 weeks
Glucose Variability assessed by 3 day SMBG | 24 weeks

SECONDARY OUTCOMES:
Target goal of HbA1c (< 7.5%) | 24 Weeks
Target goal of HbA1c (< 8.0%) | 24 Weeks
Hypoglycemia | 24 Weeks
Drug Compliance | 24 Weeks
Self monitoring blood glucose compliance | 24 Weeks
Weight change | 24 Weeks
Quality of life assessed by SF36 | 24 Weeks
Diabetes Self-Care Activities | 24 Weeks
Michigan Diabetes Knowledge Test | 24 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Soo Lim, MD, MPH, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea

REFERENCES:
- [Derived] Kim KM, Park KS, Lee HJ, Lee YH, Bae JS, Lee YJ, Choi SH, Jang HC, Lim S. Efficacy of a New Medical Information system, Ubiquitous Healthcare Service with Voice Inception Technique in Elderly Diabetic Patients. Sci Rep. 2015 Dec 11;5:18214. doi: 10.1038/srep18214. PMID 26658492